CLINICAL TRIAL: NCT00988260
Title: A Phase II Bridging Trial of Org 37462
Brief Title: Japanese Bridging Trial of Org 37462 (Study P05969)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05969
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Controlled Ovarian Stimulation
MeSH Terms: interventions — ganirelix

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ganirelix 0.125 mg (Experimental)
  Interventions: Drug: Ganirelix
- Ganirelix 0.25 mg (Experimental)
  Interventions: Drug: Ganirelix
- Ganirelix 0.5 mg (Experimental)
  Interventions: Drug: Ganirelix

INTERVENTIONS:
Drug: Ganirelix — Ganirelix 0.125 mg subcutaneous daily (SC OD) for up to 14 days
  Other Names: Org 37462; SCH 900761; Orgalutran; Ganirelix Acetate; Ganirest
  Arms: Ganirelix 0.125 mg
Drug: Ganirelix — Ganirelix 0.25 mg subcutaneous daily (SC OD) for up to 14 days
  Other Names: Org 37462; SCH 900761; Orgalutran; Ganirelix Acetate; Ganirest
  Arms: Ganirelix 0.25 mg
Drug: Ganirelix — Ganirelix 0.5 mg subcutaneous daily (SC OD) for up to 14 days
  Other Names: Org 37462; SCH 900761; Orgalutran; Ganirelix Acetate; Ganirest
  Arms: Ganirelix 0.5 mg

SUMMARY:
The purpose of this study is to find the optimal dose of Org 37462 for Japanese females undergoing controlled ovarian stimulation for in vitro fertilization intracytoplasmic sperm injection (IVF-ICSI).

ELIGIBILITY:
Inclusion Criteria:

* Japanese females of infertile married couples with an indication for COH and IVF with or without ICSI.
* At least 20 but not older than 39 years of age at the time of screening.
* A body mass index (BMI) between 18 and 29.
* Normal menstrual cycle with a range of 24-35 days and an intra-individual variation of plus or minus 3 days (but never outside the 24-35 days range).
* Infertile couple that is willing to give written informed consent.
* Determination of inclusion criteria

  * is determined in view of the planned therapeutic indication.
  * is determined based on ethical considerations for the subjects (not younger than 20) and also in view of the planned therapeutic indication (not older than 39)
  * is determined to avoid bias on the effects of Org 37462 by emaciation and obesity.
  * is determined to avoid the influences of endogenous hormones considering the purpose of this trial to select the minimal effective dose of Org 37462.
  * is determined from the ethical consideration of the subjects.

Exclusion Criteria:

* History of/or current endocrine abnormality such as polycystic ovary syndrome (PCOS) or polycystic ovaries according to USS, (treated) hyperprolactinemia or evidence of ovarian dysfunction.
* History of non- or low- ovarian response to FSH/hMG treatment.
* Abnormal cervical smear according to the Papanicolaou (>= class III) or Bethesda (>= CIN 1) scale.
* History of/or current Type I hypersensitivity (urticaria, eczema, hay fever, asthma), meaning that the subject is using prescribed medication on a regular basis or that the subjects history is prohibitive for Org 37462 treatment according to the clinical opinion of the sub-investigator.
* Any hormone value outside the reference range during the early follicular phase as measured by the central laboratory (Japan) [FSH, LH, E2, P, androstenedione (AD), dehydroepiandrosterone sulphate (DHEAS), testosterone (T), thyroid stimulating hormone (TSH) and prolactin].
* Any clinically significant abnormal laboratory value of the central laboratory (Japan) (routine hematology, blood biochemistry).
* Any ovarian and/or abdominal abnormality that would interfere with adequate ultrasound investigation of both ovaries, thus excluding subjects with only one ovary.
* Contra-indications for the use of gonadotropins i.e.,

  * tumors of ovary, breast, uterus, pituitary or hypothalamus.
  * pregnancy or lactation.
  * undiagnosed vaginal bleeding.
  * hypersensitivity to any of the substances in recFSH (FSH, sucrose, sodium citrate, polysorbate 20 and sodium chloride, L-methionine).
  * ovarian cysts or enlarged ovaries not related to PCOS.
  * malformation of the sexual organs incompatible with pregnancy.
  * fibroid tumors of the uterus incompatible with pregnancy.
* Use of hormonal preparations within 1 month prior to screening.
* Hypertension (systolic blood pressure >150 mm Hg and/or diastolic blood pressure >90 mm Hg) or treated hypertension.
* Epilepsia, diabetes, cardiovascular, gastro-intestinal, hepatic, renal, pulmonary, or abdominal disease.
* Administration of investigational drugs within 3 months prior to screening.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 266 (Actual)
Dates: Start 2003-02-03 (Actual); Primary Completion 2004-04-12 (Actual); Study Completion 2004-04-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Luteinizing Hormone (LH) rise | During treatment (1-14 days)
Intrauterine vital pregnancy rate | 5-6 weeks after embryo transfer (ET)